CLINICAL TRIAL: NCT05918575
Title: A Randomized Controlled Trial of Postextubation Use of Noninvasive Respiratory Support in Severely Obese Patients
Brief Title: Postextubation Use of Noninvasive Respiratory Support in Severely Obese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Hospital Civil de Guadalajara (Other); Medical College of Wisconsin (Other); The University of Texas Health Science Center, Houston (Other); Central DuPage Hospital (Other)
Responsible Party: Principal Investigator, Ramandeep Kaur, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23050803
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Morbid; Extubation Failure
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (NIV with HFNC) (Experimental): Patients randomized to the intervention group will receive NIV alternating with HFNC for 24 hours after extubation
  Interventions: Device: Noninvasive ventilation alternating with high flow nasal cannula
- Control Group (HFNC alone) (Active Comparator): Patients randomized to the intervention group will receive HFNC only for 24 hours after extubation
  Interventions: Device: High flow nasal cannula

INTERVENTIONS:
Device: Noninvasive ventilation alternating with high flow nasal cannula — A total of 24 hours of prophylactic respiratory support will be provided using NIV alternating with HFNC with total NIV usage of 16 hours and HFNC usage of 8 hours.
  Arms: Intervention Group (NIV with HFNC)
Device: High flow nasal cannula — A total of 24 hours of prophylactic respiratory support will be provided using HFNC alone.
  Arms: Control Group (HFNC alone)

SUMMARY:
Around 20% of the obese patients with higher body mass index (BMI) who are taken off the breathing tube and breathing machine (ventilator) end up needing it back to support breathing. The re-application of breathing tube is associated with poor outcomes, including high risk of pneumonia, longer hospital stays, and death. The purpose of this study is to assess if prophylactic use of noninvasive breathing support after removing the breathing tube lowers the chance of needing the breathing tube again.

DETAILED DESCRIPTION:
Patients with obesity are at risk of developing respiratory failure due to reduced lung volumes and chest wall compliance. Obesity is one of the easily identifiable, contributing factors of extubation failure that often leads to prolonged mechanical ventilation use and ICU stay. The early application of noninvasive respiratory support, especially NIV, has been shown to reduce reintubation rates in obese patients in a small, non-randomized study. However, prolonged use of NIV is often associated with decreased patient compliance and increased incidence of skin breakdown. HFNC is a noninvasive strategy that is comfortable, uses a nasal cannula and provides a high flow rate to meet the patient's inspiratory flow demand and thereby reduce work of breathing.

The purpose of this RCT will be to determine the effects of using NIV alternating with HFNC for reducing the treatment failure rate compared with HFNC alone in extubated patients with severe obesity. We hypothesize that early, prophylactic use of NIV alternating with HFNC will decrease the risk of respiratory failure (treatment failure) in severely obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, age ≥ 18 years old
2. Receiving invasive mechanical ventilation for ≥24 hours
3. BMI ≥40 kg/m2
4. Undergoing planned extubation per treating team
5. Arterial pH ≥7.35 or venous pH ≥ 7.31 within 30 mins of spontaneous breathing trial (SBT)

Exclusion Criteria:

1. Pregnant
2. Use of extra-corporeal membrane oxygenation
3. Chronic tracheostomy in place
4. Unplanned or accidental extubation
5. Terminal/compassionate extubation
6. Contraindication to NIV use
7. Intubated because of an acute exacerbation of COPD
8. Underlying neuromuscular disease
9. No reintubation requested by patient/family
10. Documented/known history of chronic hypercapnic respiratory failure on home NIV (including bilevel PAP).
11. Enrolled in any other outcome study
12. Treating clinician feels that HFNC or NIV are either mandatory or contraindicated for a given patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure defined by use of rescue respiratory support for acute respiratory failure in the first 72 hours after planned extubation | 72 hours
  Rescue respiratory support is defined as reintubation, use of rescue NIV or HFNC use

SECONDARY OUTCOMES:
Reintubation rate | 7 days
  Need for invasive mechanical ventilation within 7 days of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Ramandeep Kaur, PhD, Principal Investigator — Rush University Medical Center; Babak Mokhlesi, MD, Principal Investigator — Rush University Medical Center
Locations (5):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - McGovern Medical School, The University of Texas Health Science Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No